CLINICAL TRIAL: NCT06747273
Title: A Phase 1b, Multicenter, Single Dose Gene Transfer Study to Evaluate the Safety, Tolerability, and Efficacy of SRP-9004 Administered by Systemic Infusion in Limb Girdle Muscular Dystrophy Type 2D/R3 Subjects in the United States
Brief Title: Study to Evaluate the Safety, Tolerability, and Efficacy of SRP-9004 Administered by Systemic Infusion in Limb Girdle Muscular Dystrophy Type 2D/R3 Participants in the United States
Acronym: DISCOVERY
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study is being terminated due to a business decision.
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRP-9004-102
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Limb Girdle Muscular Dystrophy; Limb Girdle Muscular Dystrophy Type 2D/R3
Keywords: Limb Girdle Muscular Dystrophy Type 2D/R3; SRP-9004
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SRP-9004 (Experimental): Participants will receive a single dose of SRP-9004 on Day 1.
  Interventions: Drug: SRP-9004

INTERVENTIONS:
Drug: SRP-9004 — Intravenous (IV) infusion.

SUMMARY:
The primary objective of this study is to evaluate the safety of SRP-9004.

ELIGIBILITY:
Key Inclusion Criteria:

* Ambulatory participants, defined as able to walk without assistive aid, 10MWR <30 seconds, and NSAD total score ≥25; non-ambulatory participant, defined as 10MWR ≥30 seconds or unable to perform, and PUL 2.0 entry scale score ≥3.
* Ambulatory participants must be 4 to 20 years of age and the non-ambulatory participant must be ≥4 years of age.
* All participants must be ≤70 kilograms
* Possess 1 homozygous or 2 heterozygous pathogenic and/or likely pathogenic α-SG deoxyribonucleic acid (DNA) gene mutations as documented prior to screening.
* Able to cooperate with muscle testing.
* Participants must have adeno-associated virus (AAV) serotype Rh74 (rh74) antibody titers <1:400 (that is, not elevated) as determined by an enzyme-linked immunosorbent assay (ELISA).

Key Exclusion Criteria:

* Left ventricular ejection fraction <40% or clinical signs and/or symptoms of cardiomyopathy
* FVC ≤40% of predicted value and/or requirement for nocturnal ventilation
* Any other clinically significant illness, including neuromuscular (other than limb girdle muscular dystrophy type 2D/R3 [LGMD2D/R3]), that in the opinion of the Investigator might compromise the participant's ability to comply with the protocol required testing or procedures or compromise the participant's wellbeing, safety, or clinical interpretability.

Other inclusion/exclusion criteria apply.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs), Adverse Events of Special Interest (AESI) and Treatment-emergent Serious Adverse Events (SAEs) | Up to 60 months

SECONDARY OUTCOMES:
Change from Baseline Through Day 60 in Quantity of Alpha-sarcoglycan (α-SG) Protein Expression | Baseline, Day 60
Change from Baseline Through Month 24 in Quantity of α-SG Protein Expression | Baseline, Month 24
Change from Baseline Through Month 60 in North Star Assessment for Dysferlinopathy (NSAD) Total Score | Baseline, Month 60
Change from Baseline Through Month 60 in Performance of the Upper Limb (PUL) Version 2.0 Total Score | Baseline, Month 60
Change from Baseline Through Month 60 in Time to Rise From Floor | Baseline, Month 60
Change from Baseline Through Month 60 in Time to Ascend 4 Steps | Baseline, Month 60
Change from Baseline Through Month 60 in Time to Complete 10-meter Walk/Run (10MWR) | Baseline, Month 60
Change from Baseline Through Month 60 in Time to Complete 100-meter Walk/Run (100MWR) | Baseline, Month 60
Change from Baseline through Month 60 in Creatine Kinase (CK) Level | Baseline, Month 60
Time to Change of Disease Milestones (Loss of Ambulation) | Baseline, Month 60
Change from Baseline Through Month 60 in Skeletal Muscle Magnetic Resonance Imagining (MRI) Findings | Baseline, Month 60
Change from Baseline Through Month 60 in Wearable Device Stride Velocity 95% (SV95C) (Ambulatory Participants Only) | Baseline, Month 60
Change from Baseline Through Month 60 in Pulmonary Functions as Assessed by Forced Vital Capacity (FVC) | Baseline, Month 60
Change from Baseline Through Month 60 in Pulmonary Functions as Assessed by FVC Percentage (%) Predicted | Baseline, Month 60
Change from Baseline Through Month 60 in Pulmonary Functions as Assessed by Forced Expiratory Volume in 1 Second (FEV1) | Baseline, Month 60
Change from Baseline Through Month 60 in Pulmonary Functions as Assessed by FEV1 % Predicted | Baseline, Month 60
Change from Baseline Through Month 60 in Pulmonary Functions as Assessed by Peak Expiratory Flow Rate (PEFR) | Baseline, Month 60
Change from Baseline Through Month 60 in Pulmonary Functions as Assessed by Maximal Inspiratory Pressure (MIP) | Baseline, Month 60
Change from Baseline Through Month 60 in Pulmonary Functions as Assessed by Maximal Expiratory Pressure (MEP) | Baseline, Month 60

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of the King's Daughters, Norfolk, Virginia